CLINICAL TRIAL: NCT03369340
Title: A Single-center, Open-label, Randomized, Crossover Study to Investigate the Nicotine Pharmacokinetic Profile, Pharmacodynamics, Safety and Tolerability of Four P3P Variants in Smoking Healthy Adult Subjects
Brief Title: Nicotine Pharmacokinetics and Pharmacodynamics, Safety and Tolerability of P3P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: P3P-PK-01-CH
Record Dates: First submitted 2017-11-22; First posted 2017-12-12 (Actual); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Pharmacokinetics
Keywords: Nicotine; Nicotine-containing product

STUDY DESIGN:
Intervention Model Description: A single-center, open-label, randomized, crossover study.
Masking Description: Sponsor staff, Investigator, the subjects and the investigational site will be blinded to the randomization sequences until they are assigned. Subjects will not be informed of the complete sequence to which they have been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Product Sequence 1 (Active Comparator): Subjects will be exposed to P3P 3 on day 1 of the study, then randomized to follow a sequence of product exposure comprised of:
  P3P 2 on Day 2; P3P 4 on Day 3; P3P 1 on Day 4
  Interventions: Other: P3P 1; Other: P3P 2; Other: P3P 3; Other: P3P 4
- Product Sequence 2 (Active Comparator): Subjects will be exposed to P3P 3 on day 1 of the study, then randomized to follow a sequence of product exposure comprised of:
  P3P 4 on Day 2; P3P 1 on Day 3; P3P 2 on Day 4
  Interventions: Other: P3P 1; Other: P3P 2; Other: P3P 3; Other: P3P 4
- Product Sequence 3 (Active Comparator): Subjects will be exposed to P3P 3 on day 1 of the study, then randomized to follow a sequence of product exposure comprised of:
  P3P 1 on Day 2; P3P 2 on Day 3; P3P 4 on Day 4
  Interventions: Other: P3P 1; Other: P3P 2; Other: P3P 3; Other: P3P 4
- Product Sequence 4 (Active Comparator): Subjects will be exposed to P3P 3 on day 1 of the study, then randomized to follow a sequence of product exposure comprised of:
  P3P 1 on Day 2; P3P 4 on Day 3; P3P 2 on Day 4
  Interventions: Other: P3P 1; Other: P3P 2; Other: P3P 3; Other: P3P 4
- Product Sequence 5 (Active Comparator): Subjects will be exposed to P3P 3 on day 1 of the study, then randomized to follow a sequence of product exposure comprised of:
  P3P 2 on Day 2; P3P 1 on Day 3; P3P 4 on Day 4
  Interventions: Other: P3P 1; Other: P3P 2; Other: P3P 3; Other: P3P 4
- Product Sequence 6 (Active Comparator): Subjects will be exposed to P3P 3 on day 1 of the study, then randomized to follow a sequence of product exposure comprised of:
  P3P 4 on Day 2; P3P 2 on Day 3; P3P 1 on Day 4
  Interventions: Other: P3P 1; Other: P3P 2; Other: P3P 3; Other: P3P 4

INTERVENTIONS:
Other: P3P 1 — 2 mg of nicotine; no flavor; nicotine powder particle size of 2.25 ± 0.2 μm
Other: P3P 2 — 2 mg of nicotine; flavor; nicotine powder particle size of 2.25 ± 0.2 μm
Other: P3P 3 — 1 mg of nicotine; flavor; nicotine powder particle size of 2.25 ± 0.2 μm
Other: P3P 4 — 2 mg of nicotine; flavor; nicotine powder particle size of 1.8 ± 0.2 μm

SUMMARY:
This is a single-center, open-label, randomized, crossover study to evaluate the pharmacokinetic (PK) profiles of four P3P variants (differing in nicotine aerosol particle size, nicotine concentration and in the absence or presence of a flavoring system), following a fixed puffing regimen and an ad libitum use period. In addition, pharmacodynamic (PD) effects (subjective effects and related behavioral assessments), as well as human puffing topography, will be evaluated, to provide further insights on product safety, acceptance, and use.

DETAILED DESCRIPTION:
The goal of the proposed study is to evaluate the pharmacokinetic profiles of four P3P variants. Variants with two different nicotine contents (1 mg/product and 2 mg/product), two different nicotine aersol particle sizes and presence/absence of a flavoring system will be tested to identify which one would yield plasma nicotine concentrations as close as possible to those achieved after smoking a single cigarette. All of the subjects will initially use the lowest nicotine content product (P3P 3). Subject will continue the study using the three remaining products (P3P 1, P3P 2 and P3P 4) containing 2 mg nicotine/product in a randomly assigned sequence.

Two product use regimens: fixed puffing and ad libitum use will be applied to provide insight into nicotine absorption. The fixed puffing regimen with consistent use conditions across subjects will be applied in order to minimize variability. The 1 hour ad libitum use period will provide information on nicotine PK and product acceptance when subjects use the P3P according to their own puffing behavior which is closer to a real-world setting.

Safety and tolerability will also be assessed throughout the study.

ELIGIBILITY:
Inclusion criteria:

* Subject has signed the Informed Consent Form (ICF) and is able to understand the information provided in the ICF.
* Subject is between 21 and 65 years old.
* Subject is Caucasian.
* Smoking, healthy subject as judged by the Investigator or designee based on available assessments from the screening period.
* Subject has been smoking at least 10 commercially available cigarettes per day at least for the last 4 weeks prior to Screening Visit. Smoking status will be verified based on a urinary cotinine test (cotinine ≥ 200 ng/mL).
* Subject has been smoking for at least the last 3 years prior to Screening Visit.
* Subject does not plan to quit smoking in the next 2 months after the Screening Visit.

Exclusion criteria:

* Female subject is pregnant or breastfeeding.
* Female subject uses estrogen-containing hormonal contraception or hormone replacement therapy.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.; Milko Radicioni, MD, Principal Investigator — CROSS Research, Arzo, Ticino, Switzerland
Locations (1):
- CROSS Research, Arzo, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 subjects were screened for eligibility. 21 subjects were screen failures (10 reserve subjects were not enrolled, 9 subjects did not meet eligibility criteria, and 2 subjects withdrew.)
Pre-assignment Details: On Day 1, 19 subjects were enrolled and exposed to "P3P 3" before randomization.
  One enrolled subject withdrew after P3P 3 use before randomization. 18 subjects were randomized.
Groups:
- Product Sequence 1: Subjects will follow a sequence of product exposure comprised of:
  P3P 2 on Day 2; P3P 4 on Day 3; P3P 1 on Day 4
- Product Sequence 2: Subjects will be follow a sequence of product exposure comprised of:
  P3P 4 on Day 2; P3P 1 on Day 3; P3P 2 on Day 4
- Product Sequence 3: Subjects will follow a sequence of product exposure comprised of:
  P3P 1 on Day 2; P3P 2 on Day 3; P3P 4 on Day 4
- Product Sequence 4: Subjects will follow a sequence of product exposure comprised of:
  P3P 1 on Day 2; P3P 4 on Day 3; P3P 2 on Day 4
- Product Sequence 5: Subjects will follow a sequence of product exposure comprised of:
  P3P 2 on Day 2; P3P 1 on Day 3; P3P 4 on Day 4
- Product Sequence 6: Subjects will follow a sequence of product exposure comprised of:
  P3P 4 on Day 2; P3P 2 on Day 3; P3P 1 on Day 4
Period: Day 2
Arm/Group | Product Sequence 1 | Product Sequence 2 | Product Sequence 3 | Product Sequence 4 | Product Sequence 5 | Product Sequence 6
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Day 3
Arm/Group | Product Sequence 1 | Product Sequence 2 | Product Sequence 3 | Product Sequence 4 | Product Sequence 5 | Product Sequence 6
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Day 4
Arm/Group | Product Sequence 1 | Product Sequence 2 | Product Sequence 3 | Product Sequence 4 | Product Sequence 5 | Product Sequence 6
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Safety Population: The safety population comprised all enrolled subjects who were exposed to P3P during the study.
Arm/Group | Safety Population
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (9.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Body weight (kg) [Mean (Standard Deviation); unit: kilograms] | 72.3 (12.4)
Height (cm) [Mean (Standard Deviation); unit: centimetres] | 171 (12.6)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 24.6 (2.72)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Nicotine Concentration-time Profile
Description: To measure the plasma nicotine concentration-time profile of four P3P variants from the fixed puffing regimen, following correction of baseline nicotine levels.
Time Frame: Derived from multiple blood sampling (measured at 2 mins, 4 mins, 7 mins, 10 mins, 15 mins, 30 mins, 1 hour, 2 hours, and 4 hours post-product use) on Days 1, 2, 3 and 4
Population: Baseline correction of nicotine concentrations could be performed for 16 out of the 18 randomized subjects.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | P3P 1 | P3P 2 | P3P 3 | P3P 4
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng/mL
  2 mins after start of fixed puffing product use | 0.751 [0.447 to 1.26] | 0.336 [0.200 to 0.562] | 0.205 [0.119 to 0.351] | 0.478 [0.278 to 0.824]
  4 mins after start of fixed puffing product use | 1.56 [1.05 to 2.32] | 0.740 [0.489 to 1.12] | 0.394 [0.206 to 0.756] | 1.20 [0.762 to 1.89]
  7 mins after start of fixed puffing product use | 2.01 [1.44 to 2.79] | 1.20 [0.910 to 1.58] | 0.547 [0.330 to 0.906] | 1.66 [1.18 to 2.33]
  10 mins after start of fixed puffing product use | 2.33 [1.75 to 3.11] | 1.54 [1.23 to 1.93] | 0.701 [0.411 to 1.19] | 1.92 [1.43 to 2.57]
  15 mins after start of fixed puffing product use | 2.62 [1.92 to 3.56] | 1.78 [1.35 to 2.35] | 0.947 [0.661 to 1.36] | 2.31 [1.87 to 2.85]
  30 mins after start of fixed puffing product use | 2.40 [1.97 to 2.91] | 1.98 [1.57 to 2.51] | 0.931 [0.697 to 1.24] | 2.25 [1.91 to 2.64]
  1 hour after start of fixed puffing product use | 1.97 [1.60 to 2.42] | 1.71 [1.35 to 2.18] | 0.758 [0.573 to 1.00] | 1.85 [1.57 to 2.19]
  2 hours after start of fixed puffing product use | 1.20 [0.911 to 1.57] | 1.17 [0.897 to 1.53] | 0.383 [0.241 to 0.607] | 1.23 [1.00 to 1.51]
  4 hours after start of fixed puffing product use | 0.553 [0.391 to 0.783] | 0.568 [0.398 to 0.812] | 0.219 [0.146 to 0.329] | 0.623 [0.487 to 0.796]

2. Primary Outcome: Maximum Plasma Concentration [Cmax]
Description: To measure the maximum nicotine plasma concentration [Cmax] of four P3P variants from the fixed puffing regimen, following correction of baseline nicotine levels.
Time Frame: as for outcome 1
Population: Baseline correction of nicotine concentrations could be performed for 16 out of the 18 randomized subjects
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | P3P 1 | P3P 2 | P3P 3 | P3P 4
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng/mL | 3.08 [2.33 to 4.06] | 2.13 [1.62 to 2.81] | 1.14 [0.768 to 1.68] | 2.79 [2.10 to 3.71]

3. Primary Outcome: Time to the Maximum Nicotine Concentration [Tmax]
Description: To measure the time to maximum nicotine concentration [Tmax] of four P3P variants from the fixed puffing regimen, following correction of baseline nicotine levels.
Time Frame: as for outcome 1
Population: Baseline correction of nicotine concentrations could be performed for 16 out of the 18 randomized subjects.
Measure: Median (Full Range); unit: minutes
Arm/Group | P3P 1 | P3P 2 | P3P 3 | P3P 4
Number analyzed (Participants) | 16 | 16 | 16 | 16
minutes | 15.0 [4.00 to 60.0] | 22.5 [4.00 to 62.0] | 15.0 [4.00 to 60.0] | 15.0 [4.00 to 70.0]

4. Primary Outcome: Area Under the Concentration-time Curve From Start of Product Use (T0 Fix) to 4 Hours [AUCfix (0-4h)]
Description: To measure the area under the plasma concentration-time curve of four P3P variants from the fixed puffing regimen, following correction of baseline nicotine levels.
Time Frame: as for outcome 1
Population: Baseline correction of nicotine concentrations could be performed for 16 out of the 18 randomized subjects.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/mL*h
Arm/Group | P3P 1 | P3P 2 | P3P 3 | P3P 4
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng/mL*h | 5.84 [4.56 to 7.48] | 5.08 [3.97 to 6.50] | 2.37 [1.67 to 3.37] | 5.73 [4.45 to 7.39]

5. Secondary Outcome: Plasma Nicotine Concentration-time Profile
Description: To measure the plasma nicotine concentration-time profile of four P3P variants from the ad libitum use period, following correction of baseline nicotine levels.
Time Frame: Derived from multiple blood sampling (measured at 10 mins, 20 mins, 30 mins, 40 mins, 1 hour, 2 hours, and 4 hours during and post-ad libitum use) on Days 1, 2, 3 and 4
Population: Baseline correction of nicotine concentrations could be performed for 16 out of the 18 randomized subjects.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | P3P 1 | P3P 2 | P3P 3 | P3P 4
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng/mL
  10 minutes after start of ad libitum product use | 1.78 [1.25 to 2.53] | 1.48 [1.17 to 1.87] | 0.945 [0.647 to 1.38] | 1.49 [1.01 to 2.19]
  20 minutes after start of ad libitum product use | 2.31 [1.72 to 3.11] | 2.27 [1.69 to 3.04] | 1.21 [0.981 to 1.50] | 2.06 [1.55 to 2.74]
  30 minutes after start of ad libitum product use | 3.23 [2.63 to 3.97] | 3.17 [2.50 to 4.01] | 1.68 [1.30 to 2.17] | 2.87 [2.10 to 3.91]
  40 minutes after start of ad libitum product use | 3.96 [3.13 to 5.02] | 4.05 [3.17 to 5.17] | 1.98 [1.58 to 2.47] | 3.86 [2.88 to 5.18]
  1 hour after start of ad libitum product use | 5.28 [4.20 to 6.64] | 5.23 [4.15 to 6.58] | 2.67 [2.12 to 3.36] | 4.42 [3.26 to 5.99]
  2 hours after start of ad libitum product use | 3.91 [2.98 to 5.13] | 4.42 [3.44 to 5.69] | 1.84 [1.39 to 2.42] | 3.61 [2.66 to 4.91]
  4 hours after start of ad libitum product use | 2.07 [1.55 to 2.77] | 2.35 [1.71 to 3.22] | 0.917 [0.699 to 1.20] | 1.81 [1.38 to 2.38]

6. Secondary Outcome: Peak Plasma Nicotine Concentration [Cpeak]
Description: To measure the Peak plasma nicotine concentration [Cpeak] of four P3P variants from the ad libitum use period, following correction of baseline nicotine levels.
Time Frame: as for outcome 5
Population: Baseline correction of nicotine concentrations could be performed for 16 out of the 18 randomized subjects.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | P3P 1 | P3P 2 | P3P 3 | P3P 4
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng/mL | 5.38 [4.24 to 6.84] | 5.41 [4.26 to 6.88] | 2.63 [1.97 to 3.52] | 4.67 [3.67 to 5.95]

7. Secondary Outcome: Time to Peak Plasma Nicotine Concentration [Tpeak]
Description: To measure the time to peak plasma nicotine concentration [Tpeak] of four P3P variants from the ad libitum use period, following correction of baseline nicotine levels.
Time Frame: as for outcome 5
Population: Baseline correction of nicotine concentrations could be performed for 16 out of the 18 randomized subjects.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | P3P 1 | P3P 2 | P3P 3 | P3P 4
Number analyzed (Participants) | 16 | 16 | 16 | 16
minutes | 65.0 (22.5) | 82.4 (52.1) | 68.0 (27.2) | 61.9 (24.8)

8. Secondary Outcome: Trough Plasma Nicotine Concentration [Ctrough]
Description: To measure the trough plasma nicotine concentration [Ctrough] of four P3P variants from the ad libitum use period, following correction of baseline nicotine levels.
Time Frame: as for outcome 5
Population: Baseline correction of nicotine concentrations could be performed for 16 out of the 18 randomized subjects.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | P3P 1 | P3P 2 | P3P 3 | P3P 4
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng/mL | 1.80 [1.32 to 2.45] | 1.58 [1.16 to 2.15] | 1.13 [0.767 to 1.67] | 1.56 [1.14 to 2.13]

9. Secondary Outcome: Average of Plasma Nicotine Concentration From T0 ad Lib to 1 Hour [Caverage]
Description: To measure the average of plasma nicotine concentration [Caverage], of four P3P variants from the ad libitum use period, following correction of baseline nicotine levels
Time Frame: Derived from multiple blood sampling (measured at 10 mins, 20 mins, 30 mins, 40 mins, 1 hour during ad libitum use) on Days 1, 2, 3 and 4
Population: Baseline correction of nicotine concentrations could be performed for 16 out of the 18 randomized subjects.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | P3P 1 | P3P 2 | P3P 3 | P3P 4
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng/mL | 3.19 [2.53 to 4.02] | 3.13 [2.49 to 3.95] | 1.69 [1.29 to 2.21] | 2.87 [2.27 to 3.62]

10. Secondary Outcome: Area Under the Concentration-time Curve From Start of Product Use (T0 ad Lib) to 4 Hours [AUCad Lib (0-4h)]
Description: To measure the area under the plasma concentration-time curve of four P3P variants from the ad libitum use period, following correction of baseline nicotine levels.
Time Frame: as for outcome 5
Population: Baseline correction of nicotine concentrations could be performed for 16 out of the 18 randomized subjects.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/mL*h
Arm/Group | P3P 1 | P3P 2 | P3P 3 | P3P 4
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng/mL*h | 13.6 [10.7 to 17.3] | 14.5 [11.4 to 18.4] | 6.32 [4.73 to 8.44] | 12.1 [9.54 to 15.5]

11. Secondary Outcome: AUC of Craving for a Cigarette During and After the Fixed Puffing Regimen
Description: Measured on a Visual Analogue Scale (VAS) of 0 (no craving) to 100 (strong craving).
Time Frame: During and up to 4 hours post-product use on days 1, 2, 3 and 4
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale (millimetres)*h
Arm/Group | P3P 1 | P3P 2 | P3P 3 | P3P 4
Number analyzed (Participants) | 18 | 18 | 18 | 18
score on a scale (millimetres)*h | 40.1 [4.76 to 75.4] | 57.6 [22.3 to 92.9] | 116 [71.7 to 159] | 64.8 [29.5 to 100]

12. Secondary Outcome: AUC Craving for a Cigarette During and After the ad Libitum Use Period
Description: Measured on a Visual Analogue Scale (VAS) of 0 (no craving) to 100 (strong craving).
Time Frame: During and up to 4 hours post-product use on days 1, 2, 3 and 4
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale (millimetres)*h
Arm/Group | P3P 1 | P3P 2 | P3P 3 | P3P 4
Number analyzed (Participants) | 18 | 18 | 18 | 18
score on a scale (millimetres)*h | 76.4 [36.7 to 116] | 72.4 [32.7 to 112] | 89.6 [46.2 to 133] | 66.8 [27.2 to 107]

13. Secondary Outcome: Product Evaluation
Description: Measured with an adapted version of the modified Cigarette Evaluation Questionnaire (adapted mCEQ) following the ad libitum use period. Assessed on a 7-point scale, ranging from 1 (not at all) to 7 (extremely).
Time Frame: Within 60 minutes after the ad libitum use session on days 1, 2, 3 and 4
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | P3P 1 | P3P 2 | P3P 3 | P3P 4
Number analyzed (Participants) | 18 | 18 | 18 | 18
score on a scale
  Product Satisfaction | 3.22 [2.68 to 3.76] | 4.40 [3.86 to 4.95] | 4.42 [3.73 to 5.11] | 4.13 [3.58 to 4.67]
  Enjoyment of Respiratory Tract Sensations | 2.60 [2.04 to 3.17] | 3.88 [3.32 to 4.44] | 3.75 [3.04 to 4.46] | 3.60 [3.04 to 4.17]
  Psychological Reward | 3.12 [2.57 to 3.67] | 3.38 [2.82 to 3.93] | 3.21 [2.58 to 3.83] | 3.25 [2.70 to 3.81]
  Aversion | 1.23 [0.993 to 1.46] | 1.20 [0.965 to 1.43] | 1.10 [0.754 to 1.44] | 1.03 [0.798 to 1.27]
  Craving Reduction | 4.42 [3.78 to 5.05] | 4.58 [3.95 to 5.22] | 4.14 [3.30 to 4.98] | 4.58 [3.95 to 5.22]

14. Secondary Outcome: Sensory Parameters
Description: Measured with a Sensory Questionnaire (SQ) following the ad libitum use period. Response to each question is assessed on a 7-point scale, ranging from 1 (not at all) to 7 (extremely).
Time Frame: Within 60 minutes after the ad libitum use session on days 1, 2, 3 and 4
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | P3P 1 | P3P 2 | P3P 3 | P3P 4
Number analyzed (Participants) | 18 | 18 | 18 | 18
score on a scale
  Puffs Evaluation/Liking | 3.17 [2.64 to 3.69] | 4.22 [3.70 to 4.75] | 4.22 [3.52 to 4.93] | 3.78 [3.25 to 4.30]
  Puffs Harshness | 4.67 [4.11 to 5.23] | 3.61 [3.05 to 4.17] | 3.67 [2.87 to 4.47] | 3.72 [3.16 to 4.28]
  Puffs Similarity to Own Brand | 2.57 [1.92 to 3.23] | 2.63 [1.97 to 3.29] | 2.78 [2.01 to 3.55] | 2.30 [1.64 to 2.95]
  Puffs Strength on Tongue | 3.44 [2.67 to 4.20] | 3.10 [2.34 to 3.86] | 3.53 [2.61 to 4.44] | 2.88 [2.12 to 3.64]
  Puffs Strength in Nose | 1.89 [1.33 to 2.45] | 1.56 [0.995 to 2.12] | 1.89 [1.23 to 2.55] | 1.72 [1.16 to 2.28]
  Puffs Strength in Back of Mouth/Throat | 4.40 [3.73 to 5.07] | 3.56 [2.90 to 4.23] | 3.69 [2.78 to 4.61] | 3.79 [3.12 to 4.46]
  Puff Strength in Windpipe | 4.38 [3.72 to 5.04] | 3.44 [2.78 to 4.09] | 3.14 [2.25 to 4.02] | 3.77 [3.11 to 4.43]
  Puff Strength in Chest | 3.48 [2.75 to 4.21] | 2.81 [2.09 to 3.54] | 2.39 [1.50 to 3.28] | 3.37 [2.64 to 4.10]

15. Secondary Outcome: Human Puffing Topography (HPT) Parameters (Puff Volume) of Four P3P Variants During the Fixed Puffing Regimen Period.
Description: Descriptive statistics of total puff volume and average puff volume, of four P3P variants, during the fixed puffing regimen period.
Time Frame: During fixed puffing product use on days 1, 2, 3 and 4
Measure: Geometric Mean (95% Confidence Interval); unit: mL
Arm/Group | P3P 1 | P3P 2 | P3P 3 | P3P 4
Number analyzed (Participants) | 18 | 18 | 18 | 18
mL
  Total Puff Volume (per product) | 732 [630 to 850] | 806 [686 to 948] | 878 [714 to 1079] | 845 [733 to 975]
  Average Puff Volume (per product) | 61.0 [52.5 to 70.8] | 66.9 [56.8 to 78.8] | 72.8 [59.7 to 88.9] | 70.4 [61.1 to 81.2]

16. Secondary Outcome: Human Puffing Topography (HPT) Parameters (Puff Volume) of Four P3P Variants During the ad Libitum Use Period.
Description: Descriptive statistics of total puff volume and average puff volume, of four P3P variants, during the ad libitum use period.
Time Frame: During ad libitum product use on days 1, 2, 3 and 4
Measure: Geometric Mean (95% Confidence Interval); unit: mL
Arm/Group | P3P 1 | P3P 2 | P3P 3 | P3P 4
Number analyzed (Participants) | 18 | 18 | 18 | 18
mL
  Total Puff Volume (per product) | 1485 [1100 to 2006] | 1559 [1306 to 1861] | 1598 [1291 to 1976] | 1512 [1177 to 1941]
  Average Puff Volume (per product) | 57.5 [46.2 to 71.6] | 62.3 [51.2 to 75.9] | 65.4 [56.4 to 75.9] | 62.7 [52.5 to 74.9]

17. Secondary Outcome: Amount of Powder Aerosolized From P3P From the Fixed Puffing Regimen.
Description: Descriptive statistics of P3P weight before use, and after use, for the fixed puffing regimen.
Time Frame: Before and after fixed puffing product use on days 1, 2, 3 and 4
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | P3P 1 | P3P 2 | P3P 3 | P3P 4
Number analyzed (Participants) | 18 | 18 | 19 | 18
mg
  Weight before use | 954 (2.70) | 965 (2.11) | 966 (2.48) | 965 (2.95)
  Weight after use | 938 (6.01) | 944 (6.46) | 943 (6.46) | 942 (4.51)
  Difference of Weight (Before/After Use) | 15.6 (6.16) | 21.6 (5.89) | 22.6 (6.07) | 22.2 (3.14)

18. Secondary Outcome: Amount of Powder Aerosolized From P3P From the ad Libitum Use Period (Per Product Used).
Description: P3P weight before use, and after use, to determine the amount of powder aerosolized from P3P during Ad Libitum use (per product used).
Time Frame: Before and after ad libitum product use on days 1, 2, 3 and 4
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | P3P 1 | P3P 2 | P3P 3 | P3P 4
Number analyzed (Participants) | 18 | 18 | 19 | 18
mg
  Average Weight before use | 954 (1.83) | 964 (1.36) | 964 (1.94) | 964 (1.59)
  Average Weight after use | 937 (4.69) | 938 (4.90) | 939 (4.19) | 940 (2.28)
  Average Difference of Weight (Before/After Use) | 17.0 (4.17) | 25.9 (4.63) | 25.6 (3.92) | 23.9 (2.66)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signature of the ICF by each subject until the end of the safety follow-up period, for a duration of up to 34 days for each subject.
Groups:
- Safety Population (P3P 1): Comprising enrolled subjects who were exposed to P3P 1 during the study.
- Safety Population (P3P 2): Comprising enrolled subjects who were exposed to P3P 2 during the study.
- Safety Population (P3P 3): Comprising enrolled subjects who were exposed to P3P 3 during the study.
- Safety Population (P3P 4): Comprising enrolled subjects who were exposed to P3P 4 during the study.
Arm/Group | Safety Population (P3P 1) | Safety Population (P3P 2) | Safety Population (P3P 3) | Safety Population (P3P 4)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 4/18 | 5/18 | 4/19 | 3/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (P3P 1) (N=18) | Safety Population (P3P 2) (N=18) | Safety Population (P3P 3) (N=19) | Safety Population (P3P 4) (N=18)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocytes increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neutrophils decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specify that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT03369340/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT03369340/SAP_001.pdf